CLINICAL TRIAL: NCT00884208
Title: Fall Risk Prediction and Reduction in Community Ambulators 65 Years of Age or Older
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Guthrie Healthcare System (Other)
Responsible Party: Christy Tanton, DPT, Guthrie Healthcare System
Other Study IDs: 0903-07
Record Dates: First submitted 2009-04-17; First posted 2009-04-20 (Estimated); Last update posted 2009-04-20 (Estimated); Status verified 2009-04

CONDITIONS: Accidental Falls; Elderly; Ambulatory

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Group 1: Recommend assistive device
- Group 2: Consultation for PT assessment

SUMMARY:
The purpose of this study is to assess the diagnostic efficacy of the Tinetti Assessment, Timed up and Go test (TUG) and Gait Speed on predicting fall risk in adults 65 years of age or greater who are community ambulators.

ELIGIBILITY:
Inclusion Criteria:

* adults 65 years or older who are community ambulators.

Exclusion Criteria:

* known neurological disorder;limitation secondary to recent orthopedic condition; currently resides at skilled nursing facility

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Study Population: Adults 65 years or older who are community ambulators.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2009-04

CONTACTS AND LOCATIONS:
Overall Officials: Christy Tanton, DPT, Principal Investigator — Guthrie Healthcare System
Locations (1):
- Robert Packer Hospital, Sayre, Pennsylvania, United States